CLINICAL TRIAL: NCT06990373
Title: Establishment of Reference Intervals for Iron Test Panel for Pregnant Women at Hung Vuong Hospital
Brief Title: Iron Status of Non-anemic Pregnant Women in First Trimester
Status: Recruiting | Type: Observational
Sponsor: Hung Vuong Hospital (Other)
Responsible Party: Principal Investigator, Huan Nguyen Pham, Doctor, Hung Vuong Hospital
Other Study IDs: CS/HV/24/42
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Iron Deficiency (Without Anemia); Reference Values; Iron Deficiency Without Anemia
Keywords: NAID; IDWA; Iron deficiency; Pregnant
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With iron supplement: Pregnant women who are taking iron supplement
- Without iron supplement: Pregnant women who are not taking any iron supplement

SUMMARY:
This cross-sectional study aims to establish reference intervals for iron biomarkers-including serum iron, ferritin, total iron-binding capacity (TIBC), and transferrin saturation (TSAT)-in healthy pregnant women during the first trimester. Additionally, the study will investigate the current prevalence of non-anemic iron deficiency (NAID) in this population. By applying strict inclusion and exclusion criteria to eliminate potential confounding factors, the study seeks to provide a reliable baseline for evaluating iron status and early detection of iron deficiency without anemia among pregnant women.

DETAILED DESCRIPTION:
1. Title Reference Intervals of Iron, Ferritin, TIBC, and Transferrin Saturation in First Trimester Pregnant Women and Prevalence of Non-Anemic Iron Deficiency
2. Background and Rationale Iron deficiency (ID) is the most common micronutrient deficiency globally and a significant concern during pregnancy. Early identification of iron deficiency-even in the absence of anemia-is essential to prevent adverse maternal and fetal outcomes. However, reference intervals for iron biomarkers in early pregnancy remain inconsistent and vary across populations. Moreover, there is a paucity of data on the prevalence of non-anemic iron deficiency (NAID) during the first trimester, a critical period for fetal development. This study aims to address these gaps.
3. Objectives Primary Objective: To determine reference intervals for serum iron, ferritin, TIBC, and TSAT in healthy pregnant women during the first trimester.

   Secondary Objective: To estimate the prevalence of non-anemic iron deficiency (NAID), defined as low iron biomarkers with normal hemoglobin (Hb ≥ 11 g/dL).
4. Study Design Type: Cross-sectional observational study Setting: Antenatal care clinics at Hung Vuong Hospital, Ho Chi Minh city, Vietnam Duration: From March to June, 2025 (anticipated)
5. Study Population Inclusion Criteria

   * Pregnant women in the first trimester (gestational age ≤ 13 weeks 6 days).
   * Carrying a single live fetus.
   * Hemoglobin ≥ 11 g/dL at the time of enrollment.
   * Systolic blood pressure < 140 mmHg and diastolic < 90 mmHg.
   * Body temperature > 35°C and < 37.5°C at time of examination.
   * Attending routine antenatal care and willing to participate. Exclusion Criteria
   * History of:

   Diabetes mellitus, hypertension, hemoglobinopathies, leukemia, non-hematologic malignancies, systemic lupus erythematosus. Gastrointestinal disorders affecting iron absorption (e.g., Celiac disease, Crohn's disease, ulcerative colitis, gastric surgery).
   * Current use of acid-suppressing medications (PPIs, H2 blockers).
   * Positive screening for Treponema pallidum, HBsAg, or HIV.
   * Use of stimulants or tobacco smoking.
6. Sample Size A minimum of 120 participants is recommended for establishing reference intervals per CLSI guidelines (C28-A3), with oversampling to account for exclusions and incomplete data.
7. Data Collection Clinical Data

   * Maternal age, gestational age, BMI
   * Vital signs (BP, temperature)
   * Medical and obstetric history Laboratory Investigations
   * Hemoglobin (Hb)
   * Serum iron
   * Ferritin
   * Total iron-binding capacity (TIBC)
   * Transferrin saturation (TSAT) = (Serum iron / TIBC) × 100
8. Statistical Analysis Reference Intervals

   * Outlier detection using Dixon-Reed methods
   * Calculation of 2.5th-97.5th percentiles (non-parametric method) Prevalence of NAID
   * Defined as ferritin < 15 ng/mL or TSAT < 20% with Hb ≥ 11 g/dL (or more cutoffs to present a wide variety of prevalences of NAID). Reported as frequency and percentage with 95% confidence intervals Software
   * Statistical analysis will be performed using Jupyter Notebook (python programming language)
9. Ethical Considerations

   * Ethical approval will be obtained from the Institutional Review Board.
   * Written informed consent will be obtained from all participants.
   * Data confidentiality will be strictly maintained.
10. Significance The findings will provide local reference standards for iron parameters during early pregnancy and help clinicians better detect and manage iron deficiency before the onset of anemia. This is critical for optimizing maternal and fetal health outcomes and future study to determine best intervention for NAID patients.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending antenatal care, carrying a single live fetus.
* Systolic blood pressure at the time of examination < 140 mmHg.
* Diastolic blood pressure at the time of examination < 90 mmHg.
* Body temperature at the time of examination between >35°C and <37.5°C.
* Hemoglobin ≥ 11 g/dL

Exclusion Criteria:

* History of diabetes mellitus, hypertension, hemoglobinopathies, leukemia, non-hematologic cancers, systemic lupus erythematosus, Gastrointestinal diseases (Celiac disease, Crohn's disease and ulcerative colitis, Gastric diseases or prior gastrointestinal surgery, Irritable bowel syndrome, etc).
* Currently on gastric acid-suppressing medications: Proton pump inhibitors (e.g., Omeprazole, Lansoprazole, Esomeprazole...), H2 receptor antagonists (e.g., Ranitidine, Famotidine, Cimetidine...), Positive screening for Treponema pallidum, HBsAg, or HIV.
* Use of stimulants or tobacco smoking.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of iron supplement using women that has non-anemic iron deficiency in the first trimester | At baseline (upon enrollment)
  Non-anemic iron deficiency is defined as hemoglobin ≥ 11 g/dL and transferrin saturation (TSAT) < 20%. The prevalence will be calculated as the proportion of enrolled pregnant women meeting these criteria
Prevalence of non iron supplement using women that has non-anemic iron deficiency in the first trimester | At baseline (upon enrollment)
  Non-anemic iron deficiency is defined as hemoglobin ≥ 11 g/dL and transferrin saturation (TSAT) < 20%. The prevalence will be calculated as the proportion of enrolled pregnant women meeting these criteria
Reference Intervals for Iron Biomarkers in the First Trimester | At baseline (upon enrollment)
  Establish reference intervals (2.5th-97.5th percentile) for serum iron, ferritin, TIBC, and TSAT in healthy first-trimester pregnant women meeting inclusion criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Hung Vuong Hospital, Ho Chi Minh City, Ho Chi Minh, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Yes, the investigators plan to share individual participant data (IPD) that underlie the results reported in future publications, including de-identified data on hemoglobin, serum iron, ferritin, TIBC, transferrin saturation (TSAT), maternal demographics (age, BMI, gestational age), and relevant inclusion/exclusion criteria. Data will be available upon reasonable request for research purposes, following approval by the principal investigator and ethics board, and under a data-sharing agreement to ensure confidentiality and appropriate use.
Supporting Information: Study Protocol, CSR
Time Frame: Individual participant data will be made available beginning 6 months after publication of the main study results and will remain accessible. Data requests during this time will be reviewed and approved by the principal investigator and ethics board, subject to a data use agreement.
Access Criteria: De-identified individual participant data (IPD) will be made publicly available via a trusted data repository (e.g., Figshare) beginning 6 months after publication. No specific request or proposal is required for access. Users will be able to freely download the dataset under a standard data use license (e.g., Creative Commons Attribution [CC BY 4.0]). All shared data will be stripped of personal identifiers to protect participant confidentiality. A link to the dataset will be provided in the publication and on institutional or project websites.

REFERENCES:
- [Background] Auerbach M, Abernathy J, Juul S, Short V, Derman R. Prevalence of iron deficiency in first trimester, nonanemic pregnant women. J Matern Fetal Neonatal Med. 2021 Mar;34(6):1002-1005. doi: 10.1080/14767058.2019.1619690. Epub 2019 Jun 3. PMID 31154873
- [Background] Fisher AL, Nemeth E. Iron homeostasis during pregnancy. Am J Clin Nutr. 2017 Dec;106(Suppl 6):1567S-1574S. doi: 10.3945/ajcn.117.155812. Epub 2017 Oct 25. PMID 29070542
- [Background] Daru J, Allotey J, Pena-Rosas JP, Khan KS. Serum ferritin thresholds for the diagnosis of iron deficiency in pregnancy: a systematic review. Transfus Med. 2017 Jun;27(3):167-174. doi: 10.1111/tme.12408. Epub 2017 Apr 20. PMID 28425182
- [Background] Mei Z, Addo OY, Jefferds MED, Flores-Ayala RC, Brittenham GM. Physiologically based trimester-specific serum ferritin thresholds for iron deficiency in US pregnant women. Blood Adv. 2024 Jul 23;8(14):3745-3753. doi: 10.1182/bloodadvances.2024013460. PMID 38781318
- [Background] Pasricha SR, Tye-Din J, Muckenthaler MU, Swinkels DW. Iron deficiency. Lancet. 2021 Jan 16;397(10270):233-248. doi: 10.1016/S0140-6736(20)32594-0. Epub 2020 Dec 4. PMID 33285139